CLINICAL TRIAL: NCT06402474
Title: Effect of Two Different Surgical Positions on Pulmonary Functions in Laparoscopic Gastrectomies
Status: Active, not recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assoc. prof, Istinye University
Other Study IDs: istinye ilke
Record Dates: First submitted 2024-05-01; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Pathology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sunbed position: 30° reverse trendelenburg legs together 30° hip flexion (sunbed position)
  Interventions: Procedure: sunbed position
- control: 30° reverse trendelenburg
  Interventions: Procedure: sunbed position

INTERVENTIONS:
Procedure: sunbed position — 30° reverse trendelenburg legs together 30° hip flexion (sunbed position)

SUMMARY:
The primary purpose of the study is to investigate the effect of the 30° reverse trendelenburg position combined with the sunbed position on respiratory parameters in laparoscopic gastrectomies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who can tolerate general anesthesia and pneumoperitoneum.
* Patients who can give informed consent for surgery.
* Patients over 18 years of age
* patients with body mass index (BMI) > 30 kg/m2
* Patients with American Society of Anesthesiologists (ASA) physical status I and II

Exclusion Criteria:

* Patients with serious underlying cardiovascular disease (e.g. congestive heart failure, conduction disorders and ischemic heart disease).
* Patients with chronic kidney disease stage 3 or greater (creatinine clearance less than 60 mL/min).
* patients with a history of cerebrovascular disease such as intracranial hypertension, cerebral infarction, cerebral hemorrhage, carotid artery stenosis or cerebral ischemia;
* Patients with a history of chronic lung diseases such as chronic obstructive pulmonary disease, asthma, pulmonary bullae or respiratory failure;
* Patients who have had previous abdominal surgery, including resection of the esophagus, stomach, liver and pancreas.
* Surgeries lasting longer than 90 minutes
* Patients with ASA class IV
* patients with psychiatric disorders
* pregnant or breastfeeding patients
* patients with a history of seizures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 who underwent laparoscopic sleeve gastrectomy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-05 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
inspiratory pressure | 1 month
  effect on inspiratory pressure of two different position

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Casati A, Comotti L, Tommasino C, Leggieri C, Bignami E, Tarantino F, Torri G. Effects of pneumoperitoneum and reverse Trendelenburg position on cardiopulmonary function in morbidly obese patients receiving laparoscopic gastric banding. Eur J Anaesthesiol. 2000 May;17(5):300-5. doi: 10.1046/j.1365-2346.2000.00662.x. PMID 10926070
- [Result] Wang Y, Wang H, Wang H, Zhao X, Li S, Chen L. Exploring the intraoperative lung protective ventilation of different positive end-expiratory pressure levels during abdominal laparoscopic surgery with Trendelenburg position. Ann Transl Med. 2019 Apr;7(8):171. doi: 10.21037/atm.2019.03.45. PMID 31168452
- [Result] Shono A, Katayama N, Fujihara T, Bohm SH, Waldmann AD, Ugata K, Nikai T, Saito Y. Positive End-expiratory Pressure and Distribution of Ventilation in Pneumoperitoneum Combined with Steep Trendelenburg Position. Anesthesiology. 2020 Mar;132(3):476-490. doi: 10.1097/ALN.0000000000003062. PMID 31770148
- [Result] Mulier JP, Dillemans B, Van Cauwenberge S. Impact of the patient's body position on the intraabdominal workspace during laparoscopic surgery. Surg Endosc. 2010 Jun;24(6):1398-402. doi: 10.1007/s00464-009-0785-8. Epub 2010 Jan 7. PMID 20054583
- [Result] Gao D, Sun L, Wang N, Shi Y, Song J, Liu X, Yang Q, Su Z. Impact of 30 degrees Reserve Trendelenburg Position on Lung Function in Morbidly Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy. Front Surg. 2022 Feb 24;9:792697. doi: 10.3389/fsurg.2022.792697. eCollection 2022. PMID 35284476
- [Derived] Seyit H, Dolgun I, Bayram E, Sener FN, Cicek M. The effect of two different surgical positions on pulmonary functions in laparoscopic sleeve gastrectomies: reverse Trendelenburg vs beach chair. Surg Endosc. 2025 Mar;39(3):1829-1838. doi: 10.1007/s00464-025-11538-2. Epub 2025 Jan 21. PMID 39838149